CLINICAL TRIAL: NCT00989456
Title: Structured Patient Education in Combination With Physical Exercise as Part of the Integrated Care to Chronically Ill Patients With Chronic Obstructive Pulmonary Disease, Heart Failure and Stroke. A Randomized Controlled Intervention Trial.
Brief Title: Well Being and Rehabilitation in Chronically Ill Patients: Structured Patient Education and Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 420082351
Record Dates: First submitted 2009-09-30; First posted 2009-10-05 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Heart Failure; Stroke
Keywords: chronic obstructive pulmonary disease; Heart failure; Stroke; quality of life; self management education; physical exercise; primary health care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise and education (Experimental): Supervised physical exercise in groups, plus a self management education programme (patient education).
  Interventions: Behavioral: Self management education programme
- exercise only (Active Comparator): Supervised physical exercise in groups.
  Interventions: Behavioral: exercise only

INTERVENTIONS:
Behavioral: Self management education programme — The structured patient educational self - management programme consists of 6 weekly sessions à 2 hours. The educational programme will take place prior to one of the two weekly training sessions.
  After the initial period of 8 weeks participants are encouraged to practicing self- management on their own for a period of 9 months. They receive,in addition to standard follow - up, an offer of extra follow - up consisting of regular contact with their group supervisors in primary health care. During the last month of the intervention year educational self - management will be offered twice and focus on themes that the participants wish to refresh.
  Arms: exercise and education
Behavioral: exercise only — 6 week waiting list, followed by two weekly training sessions. After the initial period of 8 weeks participants are encouraged to practicing self- management on their own for a period of 9 months. They receive,in addition to standard follow - up, an offer of extra follow - up consisting of regular contact with their group supervisors in primary health care.
  Arms: exercise only

SUMMARY:
This study addresses self management and maintenance of health through evaluation of a program of patient education in combination with physical training and with a structured follow-up.

It is hypothesized that such a program will:

1. improve quality of life, physical functioning, coping in everyday-life
2. reduce hospitalization and (re-)admissions for patients with chronic disease, reduce consumption of home care services and can increase consumption of general practice and physiotherapy services in primary health care.
3. improve patient satisfaction and health care providers satisfaction

DETAILED DESCRIPTION:
Patients with chronically, long-lasting illness, have complex needs for treatment and care, which none of the service providers can fulfill on their own. Both patients and their relatives are in danger of experiencing severe lack of quality. Integrated care path programs are increasingly put into use. There is insufficient research-based documentation of the effect of such care paths.

The available documentation of different integrated care paths emphasizes early mobilization and discharge, rehabilitation in familiar surroundings, more effective communication and exchange of competence between the different service providers and educational self-management for patients as main elements in order to expect effect.

There are no studies that evaluate the effect of quality of life, functional skills and personal coping if group-based educational self management is combined with physical exercise and patients with different chronically illnesses participate in the same group.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age or more
* Living at home
* Capable of active participation in a group setting
* Walking distance within 550 meter in 6 minutes
* Chronic obstructive pulmonary disease (COPD) I-III
* Chronic heart disease I-III
* Stroke(0-2 on Modified Rankin Scale)

Exclusion Criteria:

* Speaking and language problems or other substantial communication problems
* Unstable medical or social situation
* Participation in another science study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | One year

SECONDARY OUTCOMES:
Sustainability of the physiological effects of muscular training (6 Minutes Walk) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Helge Garåsen, Study Director — Norwegian University of Science and Technology
Locations (5):
- Norway (5):
  - Sunndal Municipality, Sunndal, Møre Og Romsdal County
  - Surnadal municipality, Surnadal, Møre Og Romsdal County
  - Klæbu Municipality, Klæbu, Sør - Trøndelag
  - Trondheim Municipality, Trondheim, Sør Trøndelag County
  - Hitra Municipality, Hitra, Sør-Trøndelag County

REFERENCES:
- [Background] Solberg HS, Steinsbekk A, Solbjor M, Granbo R, Garasen H. Characteristics of a self-management support programme applicable in primary health care: a qualitative study of users' and health professionals' perceptions. BMC Health Serv Res. 2014 Nov 8;14:562. doi: 10.1186/s12913-014-0562-9. PMID 25380808